CLINICAL TRIAL: NCT01775943
Title: Efficacy of EGFR Tyrosine Kinase Inhibitors (EGFR TKIs) in Patients With EGFR-mutated Non-small Cell Lung Cancer Except Both Exon 19 Deletion and Exon 21 L859R: A Retrospective Analysis
Brief Title: Efficacy of EGFR TKIs in Patients With Rare EGFR-mutated NSCLC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ulsan University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Young Joo Min, Professor, Ulsan University Hospital
Other Study IDs: ISSIRES0070
Record Dates: First submitted 2013-01-18; First posted 2013-01-25 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Lung Neoplasms
Keywords: Epidermal growth factor receptor; Mutation; Lung cancer; Drug sensitivity
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Lung cancer is the leading cause of cancer-related death worldwide and is well known to remain a major health problem. Non-small-cell lung cancer (NSCLC) constitutes more than 80% of all the cases of lung cancer.

Today, NSCLC can be defined by various molecular criteria. Especially, somatic mutations within the epidermal growth factor receptor (EGFR) gene itself were discovered in a subset of NSCLC patients.

Two activating EGFR mutations are in-frame deletion in exon 19 and the substitutions for L858R in exon 21, which account for 85% of all clinically important mutations related to EGFR TKI sensitivity.

Besides two activating EGFR mutations, other EGFR mutations in NSCLC have been discovered. G719 and L861 are reported to have intermediate sensitivity to EGFR TKI. And in-frame insertions within exon 20 and T790, which are known to be resistant to EGFR TKIs.

However, there are still other EGFR mutations such as E709 and S768 as well as doublet EGFR mutations are also observed. These rare mutations have not been fully described and data on their correlation with response to EGFR-TKIs are still unclear.

Research hypothesis Rare EGFR mutations of unknown clinical significance in NSCLC patients, which are distinguish from mutations such as deletion in exon 19, L858 and insertion in exon 20, have some possibility of EGFR TKI sensitivity.

Rationale for conducting this study It has an opportunity to be shown the efficacy of EGFR TKIs in patients with rare EGFR mutation in large number of patients in Korea (Asia) during the short period.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmed non-small cell lung cancer (NSCLC), Stage IIIB or stage IV, between January 1, 2008 to December 31, 2011
2. Confirmed EGFR rare mutations (EGFR mutation except both exon 19 deletion and exon 21 L858R) using direct DNA sequencing
3. Experiences of treatment with EGFR TKIs.
4. at least one measurable and/or evaluable lesion according to RECIST criteria (version 1.1)

Exclusion Criteria:Subjects should not enter the study if any of the following exclusion criteria are fulfilled: EGFR wild type, EGFR exon 19 deletion alone, EGFR L858R alone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: comprehensive cancer hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
the efficacy of EGFR TKIs as defined by objective response rate | up to 1 year

SECONDARY OUTCOMES:
the incidence of patients with rare EGFR mutated NSCLC | up to 1 year

OTHER OUTCOMES:
the clinical characteristics of patients with rare EGFR mutated NSCLC | up to 1 year
the efficacy of EGFR TKIs as defined by disease control rate, progression-free survival and overall survival in the patients with rare EGFR mutated NSCLC | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Young Joo Min, M.D., Principal Investigator — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea